CLINICAL TRIAL: NCT02064413
Title: A Multi-Center, United States Clinical Study to Evaluate Placement Success of the ESS310 Essure® System
Brief Title: Essure (Model ESS310) Placement Rate Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 17069
Record Dates: First submitted 2014-02-14; First posted 2014-02-17 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Contraception
Keywords: Birth control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ESS310 (Experimental): All subjects that sign the informed consent and meet the eligibility criteria will be scheduled for an implant procedure.
  Interventions: Device: ESS310 (BAY1454032)

INTERVENTIONS:
Device: ESS310 (BAY1454032)

SUMMARY:
To evaluate the safety and successful placement rate of Essure Model ESS310 device and any factors that may influence the successful placement rate of this device.

ELIGIBILITY:
Inclusion Criteria:

* Females aged range 21 to 44 years
* Subjects seeking permanent contraception
* Subjects with body weight within range of 90-300 pounds (40 - 136 kilograms)
* Subjects for whom medical history indicates bilateral viable and patent fallopian tubes
* Subjects are able and willing to comply with the protocol required follow-up visits
* Subjects have fulfilled local requirements for counseling and consent to contraception and sterilization, including any required waiting periods
* Subjects provide written informed consent prior to enrolment
* Subjects who have sufficient mental capacity to understand the informed consent form (ICF), comply with the protocol requirements, and provide clinically relevant and reliable feedback regarding their experience implant and subsequent wearing of the device
* Subjects who agree that anonymized personal data will be made available to study Sponsor and requisite regional and international regulatory bodies

Exclusion Criteria:

* Subjects suspected of being or confirmed pregnant
* Subjects post-partum or undergone pregnancy termination ≤6 weeks of scheduled insert placement
* Subjects who have known proximal tubal occlusion in either fallopian tube
* Subjects who have undergone fallopian tube sterilization procedure
* Subjects who have had total or partial salpingectomies
* Subjects diagnosed with tubal, endometrial, or myometrial pathology which may prevent fallopian tube ostia access
* Subjects diagnosed with unicornuate uterus
* Subjects diagnosed with active or currently being treated upper or lower pelvic infection
* Subjects with gynecologic malignancy
* Subjects who are currently taking corticosteroids
* Subjects with a known allergy to all contrast media available for use in HSG (Hysterosalpingogram)
* Subjects scheduled to undergo concomitant intrauterine procedures at the time of insert placement (e.g., endometrial ablation, fibroid resection by hysteroscopy, endometrial polypectomy). Intrauterine device removal is not considered a concomitant procedure.
* Subjects with any general health condition or systemic disease that may represent, in the opinion of the physician, a potential increased risk associated with device use or pregnancy
* Subjects with a close affiliation with the investigational site, e.g. closely related or affiliated with the investigator (such as dependent, employee or student of the investigational site, or sponsor's staff)

Ages: 21 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 134 (Actual)
Dates: Start 2014-03-17 (Actual); Primary Completion 2014-10-02 (Actual); Study Completion 2014-11-26 (Actual)

PRIMARY OUTCOMES:
Rate of successful bilateral placement of the ESS310 insert at first attempt in subjects who undergo attempted ESS310 placement | Day 1

SECONDARY OUTCOMES:
Successful bilateral placement rate of the ESS310 insert at first attempt in all subjects who undergo hysteroscopy with the intent of having bilateral ESS310 placement | Day 1
Evaluation of investigator questionnaire regarding ESS310 design and usability | Day 1
  Potential aspects of the ESS310 design and usability that may impact bilateral placement rate at first attempt
Evaluation of investigator questionnaire regarding potential factors predictive of failure to achieve bilateral placement of the ESS310 insert at first attempt | Day 1
Hysteroscopy time to perform the procedure | Day 1
Number of participants with Adverse device effects (ADE) as a measure of safety and tolerability | 1 week
Number of participants with Adverse procedure-related events as a measure of safety and tolerability | Day 1, 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (16):
- United States (16):
  - Glendale, Arizona
  - Phoenix, Arizona
  - Colorado Springs, Colorado
  - Augusta, Georgia
  - Fort Wayne, Indiana
  - Newburgh, Indiana
  - Grand Blanc, Michigan
  - Saginaw, Michigan
  - Wayne State University Physicians Group, Southfield, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Winston-Salem, North Carolina
  - Dayton, Ohio
  - Tennessee Women's Care, PC, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Fort Worth, Texas
  - Houston, Texas